CLINICAL TRIAL: NCT00944606
Title: Vitamin D vs Placebo in the Treatment of Vague Musculoskeletal Pain in Children
Brief Title: Vitamin D Versus Placebo in the Treatment of Vague Musculoskeletal Pain in Children
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: inability to recruit subjects
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Elizabeth Szalay, Professor, Pediatric Orthopaedics & Pediatrics, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HRRC 09-167
Record Dates: First submitted 2009-07-21; First posted 2009-07-23 (Estimated); Last update posted 2012-03-01 (Estimated); Status verified 2012-02

CONDITIONS: Hypovitaminosis D
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D (Active Comparator)
  Interventions: Dietary Supplement: Vitamin D
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo candy

INTERVENTIONS:
Dietary Supplement: Vitamin D — 2000-3000 IU Vitamin D daily x 6 weeks
  Other Names: Rainbow Light
  Arms: Vitamin D
Other: Placebo candy — candy gum drops
  Arms: Placebo

SUMMARY:
Other studies suggest that low Vitamin D levels may contribute to musculoskeletal pain.

Hypothesis: Administration of oral Vitamin D supplements will improve vague musculoskeletal pain in children.

ELIGIBILITY:
Inclusion Criteria:

* ages 5-14
* healthy
* vague musculoskeletal pain without diagnosis

Exclusion Criteria:

* medications (steroids, seizure medications, birth control pills or shot)
* endocrinopathies

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2009-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Lessening of musculoskeletal pain level and frequency | 6 weeks

SECONDARY OUTCOMES:
Improvement of serum 25 OH Vitamin D level | 6 weeks
Decline of serum parathyroid hormone levels | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Szalay, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico General Clinical Research Center, Albuquerque, New Mexico, United States